CLINICAL TRIAL: NCT01282268
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of STX209 (Arbaclofen) Administered for the Treatment of Social Function in Adolescents and Adults With Fragile X Syndrome
Brief Title: Efficacy and Safety Study of STX209 (Arbaclofen) for Social Withdrawal in Adolescents and Adults With Fragile X Syndrome
Acronym: Harbor-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 209FX301
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Fragile X Syndrome
Keywords: fragile X syndrome; autism spectrum disorder
MeSH Terms: conditions — Fragile X Syndrome; Autism Spectrum Disorder | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arbaclofen (Active Comparator)
  Interventions: Drug: arbaclofen
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: arbaclofen — orally disintegrating tablet
  Other Names: STX209
  Arms: Arbaclofen
Drug: placebo — orally disintegrating tablet
  Arms: Placebo

SUMMARY:
To explore the efficacy, safety and tolerability of STX209 (arbaclofen) administered for the treatment of social withdrawal in adolescents and adults with fragile X syndrome (FXS)

ELIGIBILITY:
Inclusion Criteria:

* Molecular documentation of the full FMR1 mutation
* Current pharmacological treatment regimen has been stable for at least 4 weeks prior to Screening.
* Subjects with a history of seizure disorder must currently be receiving treatment with antiepileptics and must have been seizure free for 6 months, or must be seizure free for 3 years if not currently receiving antiepileptics.
* If the subject is already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, participation in these programs must have been continuous during the 2 months prior to Screening

Exclusion Criteria:

* Subjects with any condition, including alcohol and drug abuse, which might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being.
* Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Subjects who have taken another investigational drug within the last 30 days.
* Subjects who are not able to take oral medications.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist - FXS Social Avoidance Subscale | At 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, M.D., Study Director — Seaside Therapeutics, Inc.
Locations (24):
- United States (24):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Miller Children's Hospital Research Administration, Long Beach, California
  - University of California-Davis, M.I.N.D. Institute, Sacramento, California
  - Psychiatric Centers at San Diego, San Diego, California
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - University of Miami, Mailman Center for Child Development, Miami, Florida
  - Lake Mary Pediatrics, Orange City, Florida
  - Emory University School of Medicine, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - University of Missouri, Thompson Research Center for Autism & Neurodevelpmental Disorders, Columbia, Missouri
  - Seaver Autism Center, Mount Sinai Medical Center, New York, New York
  - New York State Institute for Basic Research in Developmental Disabilities, Staten Island, New York
  - Duke University Clinical Research Unit, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - University of Oklahoma, Physician's Child Study Center, Oklahoma City, Oklahoma
  - Suburban Research Associates/Elwyn Genetics, Media, Pennsylvania
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Red Oaks Psychiatry Associates, P.A., Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington